CLINICAL TRIAL: NCT00471536
Title: A Phase II Safety and Efficacy Study With the VEGF Receptor Tyrosine Kinase Inhibitor GW786034 in Patients With Metastatic Urothelial Cancer
Brief Title: Pazopanib in Treating Patients With Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00203; NCI-2009-00203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000543460; MAYO-MC0553; MC0553 (Other: Mayo Clinic); 7661 (Other: CTEP); N01CM62205 (NIH)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2013-12

CONDITIONS: Distal Urethral Cancer; Proximal Urethral Cancer; Recurrent Bladder Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder; Urethral Cancer Associated With Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — pazopanib

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive 800 mg oral pazopanib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pazopanib hydrochloride

INTERVENTIONS:
Drug: pazopanib hydrochloride — 800 mg Given orally
  Other Names: GW786034B; Votrient

SUMMARY:
This phase II trial is studying the side effects and how well pazopanib works in treating patients with metastatic urothelial cancer. Pazopanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the anti tumor activity and toxicity profile of pazopanib hydrochloride in patients with metastatic urothelial cancer.

SECONDARY OBJECTIVES:

I. Evaluate the pharmacokinetics of pazopanib hydrochloride in these patients. II. Evaluate pre- and post-treatment changes in circulating endothelial cells, monocytes and platelets, and angiogenesis-related factors in these patients.

OUTLINE: This is a multicenter study. Patients receive oral pazopanib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically for correlative studies and pharmacological studies. Samples are analyzed for vascular endothelial growth factor (VEGF) and soluble VEGF receptor II concentration via ELISA. Circulating endothelial cells are also measured.

After completion of study treatment, patients are followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed transitional cell cancer of the urothelium or bladder

  * Metastatic disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan
* No known brain metastases
* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* PT/INR/PTT ≤ 1.2 times ULN
* No proteinuria > 1+ on two consecutive dipsticks measured ≥ 1 week apart
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to pazopanib hydrochloride or other agents used in the study
* No condition that impairs the ability to swallow and retain pazopanib hydrochloride tablets, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication
  * Requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No uncontrolled illness that would limit compliance with study therapy including, but not limited to, any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situations
* No QTc prolongation (defined as a QTc interval ≥ 480 msecs) or other significant ECG abnormalities (e.g., frequent ventricular ectopy, evidence of ongoing myocardial ischemia)
* No other conditions, including any of the following:

  * Serious or non-healing wound, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
  * Cerebrovascular accident within the past 6 months
  * Myocardial infarction, cardiac arrhythmia, or admission for unstable angina within the past 12 weeks
  * Venous thrombosis within the past 12 weeks
  * New York Heart Association (NYHA) class III or IV heart failure

    * Asymptomatic NYHA class II heart failure on treatment allowed
* No other active second malignancy other than non-melanoma skin cancer

  * Patients are not considered to have an active malignancy if they have completed anti-cancer therapy and are considered by their physician to be ≤ 30% risk of relapse
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 4 weeks since prior radiotherapy
* Prior palliative radiotherapy to metastatic lesions allowed provided there is ≥ 1 measurable and/or evaluable lesion(s) that has not been irradiated
* At least 4 weeks since prior surgery
* One prior chemotherapy regimen for metastatic urothelial or bladder cancer
* More than 12 weeks since prior cardiac angioplasty or stenting
* Prior adjuvant or neoadjuvant therapy allowed
* No prior experimental treatment for metastatic disease
* No other prior or concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent CYP2C9 substrates, including any of the following:

  * Anticoagulants (e.g., warfarin [therapeutic doses only])

    * Low molecular weight heparin and prophylactic low-dose warfarin (≤ 2 mg daily) allowed
  * Oral hypoglycemics (e.g., glipizide, glyburide, tolbutamide, glimepiride, or nateglinide)
  * Ergot derivatives (e.g., dihydroergotamine, ergonovine, ergotamine, or methylergonovine)
  * Antipsychotics (e.g., pimozide or clozapine)
  * Erectile dysfunction agents (e.g., sildenafil, tadalafil, or vardenafil)
  * Antiarrhythmics (e.g., bepridil, flecainide, lidocaine, mexiletine, amiodarone, quinidine, or propafenone)
  * Immune modulators (e.g., cyclosporine, tacrolimus, or sirolimus)
  * Miscellaneous drugs (e.g., theophylline, quetiapine, risperidone, tacrine, or atomoxetine)
* No other concurrent anticancer agents or therapies
* No concurrent medications that are associated with a risk of QTc prolongation and/or Torsades de Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka Vaishampayan, Principal Investigator — Mayo Clinic
Locations (9):
- United States (7):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Cox Medical Center, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong, China
- Gangnam Severance Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nineteen participants were accrued between October 2008 and December 2009.
Pre-assignment Details: Of the 19 participants accrued, one participant canceled prior to treatment evaluation, and therefore was excluded from toxicity analysis. This participant was included in the primary endpoint analysis.
Groups:
- Treatment (Enzyme Inhibitor Therapy): Patients receive oral pazopanib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 19
Completed | 18
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 66 [42 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 14
  Korea, Republic of | 1
  Hong Kong | 2
  Australia | 2

OUTCOME MEASURES:

1. Primary Outcome: Best Tumor Response (Complete [CR] or Partial Response [PR] by Response Evaluation Criteria in Solid Tumors [RECIST])
Description: Tumor response is defined as the total number of eligible patients whose disease has a complete or partial response to GW786034 according to the RECIST criteria. Per RECIST v1.0 criteria:
  A Complete Response (CR) requires the disappearance of all target lesions.
  A Partial Response (PR) requires >=30% decrease in the sum of the longest diameter of target lesions from baseline measurement.
  All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response.
Time Frame: Participants will be evaluated every 8 weeks during treatment and up to 1 year after completion of treatment.
Population: All participants meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluated for response.
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 19
participants
  Partial Response (PR) | 0
  Complete Response (CR) | 0

2. Secondary Outcome: Adverse Events Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: The maximum grade for each adverse event considered to be at least possibly related to treatment will be recorded. Frequency tables will be constructed.
Time Frame: Every 4 weeks during treatment (maximum duration was 44 weeks)
Population: Eighteen of the 19 participants accrued to the study were evaluable for adverse events.
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
participants
  Grade 3 Adverse Events | 7
  Grade 4 or Higher Adverse Events | 0

3. Secondary Outcome: Confirmed Tumor Response (CR and PR)
Description: Tumor response is defined as the total number of eligible patients whose disease has a complete or partial response to GW786034 according to the RECIST criteria. A confirmed response is defined as a CR or PR and is documented on 2 consecutive evaluations.
Time Frame: Documented on 2 consecutive evaluations 8 weeks apart from the start of the treatment until disease progression/recurrence, assessed up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 19
participants
  Confirmed Partial Response (PR) | 0
  Confirmed Complete Response (CR) | 0

4. Secondary Outcome: Duration of Response
Description: The distribution of response durations will be estimated using the Kaplan-Meier method.
Time Frame: From the time an objective response is first noted to be either a CR or PR to the date progression is documented, assessed up to 1 year
Population: There were no responses.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Disease Progression
Description: The distribution of progression-free survival times will be estimated using the Kaplan-Meier method.
Time Frame: Every 3 months from registration until progressive disease (PD), assessed up to 2 years after registration
Population: All participants were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 19
months | 1.85 [1.77 to 3.71]

6. Secondary Outcome: Survival Time
Description: The distribution of survival times will be estimated using the Kaplan-Meier method.
Time Frame: Time from registration until death due to any cause, assessed every 6 months after PD for up to 2 years after registration
Population: all participants were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 19
months | 5.83 [3.38 to 7.98]

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=18)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=18)
Hemoglobin decreased (Blood and lymphatic system disorders) | 13 (32)
Flashing vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (7)
Anal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 9 (17)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (3)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 10 (23)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (12)
Fatigue (General disorders) | 17 (53)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Urostomy site bleeding (Injury, poisoning and procedural complications) | 1 (5)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (11)
Bilirubin increased (Investigations) | 2 (2)
Leukocyte count decreased (Investigations) | 8 (15)
Lymphocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 3 (6)
Platelet count decreased (Investigations) | 10 (19)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (19)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Taste alteration (Nervous system disorders) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 7 (20)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (6)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 4 (9)
Hypertension (Vascular disorders) | 9 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less